CLINICAL TRIAL: NCT05730192
Title: Evaluation of Artificial Intelligence for Detection of Gastrointestinal Lesions in Endoscopy (EAGLE)
Brief Title: EAGLE Trial CADDIE Artificial Intelligence Endoscopy
Acronym: EAGLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odin Medical (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RCT-2022-01
Record Dates: First submitted 2023-01-23; First posted 2023-02-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Polyp of Colon; Adenoma Colon
Keywords: Screening; Surveillance; Artificial Intelligence; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: Parallel trial design
Who Masked: Outcomes Assessor
Masking Description: Histology of the polyps is performed by the pathologist blinded to the study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CADDIE colonoscopy (CADDIE Arm) (Experimental): CADDIE is a computer-assisted detection (CADe) device used in conjunction with endoscopy for the detection of abnormal lesions in the gastrointestinal tract.
  Interventions: Device: CADDIE
- Standard high-definition white light colonoscopy (Control Arm) (Active Comparator): Patients will receive a standard colonoscopy
  Interventions: Device: CADDIE

INTERVENTIONS:
Device: CADDIE — A colonoscopy is an examination of the bowels using a colonoscope, or a thin, flexible tube with a light and camera. It can help identify issues like colorectal cancer, polyps, and ulcers.
  Other Names: Colonoscopy

SUMMARY:
The EAGLE study is a prospective randomized controlled multicenter parallel design trial, for the assessment of clinical performance of the CADDIE device and to confirm that the device performs as expected.

DETAILED DESCRIPTION:
The EAGLE study will be conducted with a parallel design. Patients who meet the study inclusion/exclusion criteria will be randomized in a 1:1 ratio to receive either computer-aided colonoscopy (CADDIE Arm) using CADDIE or standard colonoscopy without CADe (Control Arm). All resected polyps will be submitted for histologic examination.

ELIGIBILITY:
Inclusion Criteria:

1. Screening or surveillance colonoscopy
2. Age 40 years or older
3. Informed consent

Exclusion Criteria:

1. Emergency colonoscopies
2. Inflammatory bowel disease (IBD)
3. Colorectal Cancer (CRC)
4. Previous Colorectal Cancer (CRC)
5. Previous colonic resection
6. Returning for a planned elective therapeutic colonoscopy.
7. Polyposis syndromes (familial adenomatous polyposis)
8. Contraindication for biopsy or polypectomy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 985 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Number of Adenoma per colonoscopy (APC) | During the procedure/surgery
  Superiority of CADDIE Arm vs. control.
Positive percent agreement (PPA) | During the procedure/surgery
  Non inferiority of CADDIE Arm vs. control.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, Prof., Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (9):
- Israeli-Georgian Medical Research Clinic Healthycore, Tbilisi, Georgia
- Sana Klinikum Lichtenberg, Berlin, Germany
- Italy (3):
  - Humanitas Mater Domini, Castellanza, Varese
  - Humanitas Catania, Catania
  - Humanitas Research Hospital, Milan
- Poland (3):
  - H-T. Centrum Medyczne, Tychy
  - The Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
  - Przychodnia Polskiej Fundacji Gastroenterologii, Warsaw
- University Hospital "Clinico Lozano Blesa" of Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kader R, Hassan C, Lanas A, Romanczyk M, Romanczyk T, Kotowski B, Homedes CS, Mangiavillano B, Bonanno G, Lovat LB, Kaminski M, Faiss S, Repici A. A novel cloud-based artificial intelligence for real-time detection of colorectal neoplasia - a randomized controlled trial (EAGLE). NPJ Digit Med. 2025 Dec 26;9(1):84. doi: 10.1038/s41746-025-02270-1. PMID 41449203
- See also: Meditrial Clinical Research Organization — https://www.meditrial.net/
- See also: Odin Vision Cloud Connected Endoscopy — https://odin-vision.com/